CLINICAL TRIAL: NCT03327909
Title: Timing of Antihypertensive Medications on Key Outcomes in Hemodialysis
Acronym: TAKE-HOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Satellite Healthcare (Other)
Responsible Party: Principal Investigator, Tara I-Hsin Chang, Assistant Professor of Medicine (Nephrology), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAKE-HOLD
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: ESRD; Hemodialysis Complication; Blood Pressure
Keywords: Intradialytic Hypotension, Hypertension, Ambulatory Blood Pressure
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension

STUDY DESIGN:
Intervention Model Description: Cluster randomized parallel group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAKE (Experimental): Participants in TAKE units will be advised to take all antihypertensive medications as prescribed, including on the morning of dialysis.
  Interventions: Behavioral: TAKE vs. HOLD
- HOLD (Experimental): Participants in the HOLD units will advised to hold the dose of the antihypertensive medications prior to the dialysis session on the morning of the dialysis days. Participants can choose whether they wish to take the antihypertensive medication that was held at any time after the dialysis session has ended.
  Interventions: Behavioral: TAKE vs. HOLD

INTERVENTIONS:
Behavioral: TAKE vs. HOLD — All participants will be told to take once daily antihypertensive medications at night. Timing of other antihypertensive medication administration will differ depending on whether the participant is randomized to the TAKE or HOLD arm.

SUMMARY:
For patients with kidney failure requiring hemodialysis treatment, sometimes the blood pressure will drop too low during dialysis. In an effort to prevent that from occurring, patients are frequently told to skip doses of their blood pressure medications. However, whether this actually prevents blood pressure drops during dialysis, and whether it may cause more uncontrolled high blood pressure is unknown. TAKE-HOLD will study the effect of taking or holding blood pressure medication on blood pressure for patients on hemodialysis.

DETAILED DESCRIPTION:
High blood pressure (BP) is a major modifiable risk factor for cardiovascular disease, and upwards of 90% of patients with end- stage renal disease (ESRD) have high BP. Appropriate BP management, therefore, is a fundamental part of patient care in ESRD, yet the question of when best to take antihypertensive medications relative to the hemodialysis treatment session remains unanswered. Many patients on hemodialysis suffer from an abrupt fall in BP during the dialysis session (i.e., intradialytic hypotension [IDH]), a phenomenon that is associated with numerous adverse outcomes. In an attempt to minimize IDH, patients are often told to withhold antihypertensive medications prior to hemodialysis, and current guidelines suggest taking antihypertensive medications at night to minimize IDH. However, there are no data regarding the safety of these antihypertensive medication timing strategies, or whether these strategies are effective in reducing IDH.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. On in-center thrice weekly hemodialysis
3. Dialysis start time in the morning
4. Taking at least one antihypertensive medication

Exclusion Criteria:

1. Initiation of hemodialysis within previous 90 days
2. Inability to provide informed consent
3. Currently participating in another clinical trial (intervention study)
4. >2 unexcused missed dialysis sessions in the previous 30 days
5. Documented heart failure with reduced ejection fraction (left ventricular ejection fraction < 40%)
6. Cardiovascular event (e.g. myocardial infarction, stroke, heart failure) or procedure (e.g., coronary artery bypass, peripheral arterial bypass grafting, carotid artery procedures, aortic procedures) or hospitalization for unstable angina within the previous 90 days
7. End-stage liver disease
8. Planned kidney transplant within the next 90 days
9. Planned dialysis modality switch (to home hemodialysis, peritoneal dialysis, nocturnal hemodialysis) within the next 90 days
10. Pregnancy, currently trying to become pregnant
11. Active infection requiring antibiotic, antifungal or antiviral therapies
12. Any factors judged by the treatment team to be likely to limit adherence to the interventions

    1. Active alcohol or substance abuse within the last 12 months
    2. Plans to move outside of the treatment area within in the next 90 days
    3. Other medical, psychiatric, or behavioral factors that in the judgement of the study team may interfere with study participation or the ability to follow the intervention protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Intradialytic Hypotension | 4-week intervention period
  Number of participants with ≥30% of dialysis sessions with symptomatic or asymptomatic IDH.

SECONDARY OUTCOMES:
Poorly controlled pre-dialysis blood pressure | 4-week intervention period
  Number of participants with ≥30% of dialysis sessions with pre-dialysis systolic BP > 160 mm Hg
Dialysis Tolerability | 4-week intervention period
  Number of participants with ≥30% of dialysis sessions with post-dialysis weight > prescribed dry weight or delivered length of dialysis < prescribed length. We will also assess dialysis symptoms using the Dialysis Symptom Index.

OTHER OUTCOMES:
44-hour ambulatory blood pressure | Final week of the 4-week intervention period
  Compare the number of hours spent in the desired systolic BP range of 110-150 mm Hg in patients in TAKE versus HOLD units. We will also compare the number of patients who demonstrate nocturnal dipping patterns of BP in the TAKE and HOLD units.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Satellite Health Care, Menlo Park, California
  - Satellite Health Care, San Carlos, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang TI, Tatoian ET, Montez-Rath ME, Chertow GM. Timing of Antihypertensive Medications on Key Outcomes in Hemodialysis: A Cluster Randomized Trial. Kidney360. 2021 Sep 16;2(11):1752-1760. doi: 10.34067/KID.0001922021. eCollection 2021 Nov 25. PMID 35373003